CLINICAL TRIAL: NCT07361965
Title: Validity and Reliability of the Mixed Reality-Based Adaptation of the Timed Up and Go, Five-Repetition Sit-to-Stand, and 25-Foot Walk Tests in Individuals With Multiple Sclerosis
Brief Title: Validity and Reliability of Mixed Reality-Based Mobility Tests in Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_MS_MR_ADAPTATION
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Mixed Reality
Keywords: Multiple Sclerosis; Mixed Reality; Functional Mobility; Validity; Reliability; Digital Assessment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Multiple Sclerosis: Individuals with multiple sclerosis aged 18-60 years.
  Interventions: Other: Clinical Assessments

INTERVENTIONS:
Other: Clinical Assessments — Participants with multiple sclerosis will undergo EDSS assessment, functional mobility tests (TUG, 5xSTS, and T25FW; conventional and mixed reality-based), fatigue (MFIS), walking performance (MSWS-12), knee extensor muscle strength, handgrip strength, and participant satisfaction evaluations. Conventional tests will be performed prior to mixed reality-based assessments; MR-based tests will be conducted using the Meta Quest 3 and repeated one week later for test-retest reliability.

SUMMARY:
Multiple sclerosis (MS) is a demyelinating and neurodegenerative disease of the central nervous system, with common symptoms including muscle weakness, balance impairments, gait difficulties, and fatigue. These symptoms significantly affect individuals' functional mobility, independence, and quality of life. In individuals with MS, reduced lower extremity muscle strength leads to decreased walking speed and loss of balance, resulting in substantial limitations in activities of daily living.

Conventional clinical assessment tools, such as the Timed Up and Go (TUG), Five-Repetition Sit-to-Stand Test (5xSTS), and the Timed 25-Foot Walk (T25FW), have been widely used for many years to evaluate functional mobility in individuals with MS. However, these tests typically rely on unidimensional measurement parameters and may demonstrate subjective variability depending on the testing environment and the examiner's experience. Advances in measurement technologies now allow these clinical tests to be transformed into more objective, standardized, and interactive assessment tools.

Virtual reality (VR) provides a new perspective for the assessment of motor performance by enabling three-dimensional and interactive simulations of real-world scenarios. VR-based applications allow for the simultaneous evaluation of both motor and cognitive components while also increasing individuals' motivation and engagement. Previous studies have demonstrated that VR technology is effective in neurological rehabilitation, particularly in improving balance, walking speed, and functional mobility in the MS population. In contrast to VR, mixed reality (MR) is a technology that allows individuals to maintain interaction with the real environment while integrating virtual objects into the physical space.

The existing literature reveals a notable gap in research focusing on the validity and reliability of VR or MR-based functional tests in individuals with multiple sclerosis. However, no studies to date have investigated the adaptation of lower extremity functional tests (TUG, 5xSTS, and T25FW) to a mixed reality environment. Therefore, the primary rationale of this study is to evaluate the digital applicability of commonly used functional tests in individuals with MS on the Meta Quest 3 virtual reality platform and to determine the validity and reliability of these tests. Additionally, this study aims to examine the relationships between data obtained from the virtual tests and fatigue (Modified Fatigue Impact Scale, MFIS), walking performance (12-Item Multiple Sclerosis Walking Scale: MSWS-12), and knee extensor muscle strength in order to establish the convergent validity of this novel approach.

The findings of this study are expected to contribute to the development of an objective, standardized, safe, and innovative digital assessment tool for functional evaluation in individuals with multiple sclerosis. Furthermore, the results will strengthen the scientific foundation for remote monitoring of the rehabilitation process and for the development of personalized treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of multiple sclerosis (MS) established by a neurologist,
* Not being in a relapse phase and having no MS relapse within the past 6 months,
* Aged between 18 and 60 years,
* Disease severity within an Expanded Disability Status Scale (EDSS) range of 1-5 (mild to moderate functional impairment),
* Visual, auditory, and vestibular functions sufficient to tolerate mixed reality-based applications,
* Adequate cognitive capacity to actively participate in the study (e.g., Mini-Mental State Examination score ≥ 24),
* Ability to read, understand, and follow instructions in Turkish,
* Willingness to participate voluntarily in the study and provision of written informed consent.

Exclusion Criteria:

* Having experienced a multiple sclerosis relapse or undergone a change in MS-related treatment within the past 6 months,
* Presence of severe musculoskeletal disorders (e.g., fracture, arthritis, advanced osteoarthritis, muscle tear) that may interfere with test performance,
* Presence of severe cardiopulmonary disease (e.g., uncontrolled hypertension, heart failure, chronic obstructive pulmonary disease) or any medical condition that may pose a risk during exercise testing,
* Risk of loss of balance or spatial disorientation in the mixed reality environment due to visual, vestibular, or auditory impairments,
* Inability to perform functional tests due to severe spasticity, contractures, or orthopedic deformities,
* History of epilepsy, migraine, or other neurological conditions that contraindicate the use of mixed reality or virtual reality devices,
* Inability to understand test instructions due to cognitive impairment or severe mental health disorders (e.g., dementia, major depression, psychotic disorders),
* Experiencing dizziness, nausea, or virtual reality-related symptoms (VR sickness) during testing,
* Insufficient motivation or poor compliance that may hinder participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with MS who applied to the Selçuk University Faculty of Medicine Hospital MS Living Center
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test - Mixed Reality (TUG-MR) | Baseline and 1-week follow-up
  This outcome measure will be used to assess functional mobility, balance, and lower extremity performance in individuals with multiple sclerosis using a mixed reality-based digital adaptation of the Timed Up and Go test. Test completion time will be automatically recorded by the system.
Five-Repetition Sit-to-Stand Test - Mixed Reality (5xSTS-MR) | Baseline and 1-week follow-up
  This outcome measure will be used to assess lower extremity muscle strength and functional mobility using a mixed reality-based adaptation of the Five-Repetition Sit-to-Stand test. Test duration will be automatically recorded.
Timed 25-Foot Walk - Mixed Reality (T25FW-MR) | Baseline and 1-week follow-up
  This outcome measure will be used to assess walking speed and functional mobility in individuals with multiple sclerosis using a mixed reality-based version of the Timed 25-Foot Walk test. Test time will be automatically recorded by the system.

SECONDARY OUTCOMES:
Timed Up and Go Test - Conventional | Baseline
  The conventional Timed Up and Go test will be administered to assess functional mobility and balance. This test is a valid and reliable clinical measure in individuals with multiple sclerosis.
Five-Repetition Sit-to-Stand Test - Conventional | Baseline
  The conventional Five-Repetition Sit-to-Stand test will be used to assess lower extremity muscle strength and functional mobility.
Timed 25-Foot Walk - Conventional | Baseline
  The conventional Timed 25-Foot Walk test will be administered to assess walking speed and mobility. This test is a component of the Multiple Sclerosis Functional Composite.
Expanded Disability Status Scale (EDSS) | Baseline
  This scale will be administered by a physician to determine the level of neurological disability in individuals with multiple sclerosis.
Modified Fatigue Impact Scale (MFIS) | Baseline
  This scale will be used to assess the impact of fatigue on physical, cognitive, and psychosocial functioning in individuals with multiple sclerosis.
Multiple Sclerosis Walking Scale-12 (MSWS-12) | Baseline
  This self-reported questionnaire will be used to assess walking performance and the impact of walking difficulties on daily life in individuals with multiple sclerosis.
Knee Extensor Muscle Strength | Baseline
  Knee extensor muscle strength will be measured using a handheld digital dynamometer to assess lower extremity muscle strength.
Handgrip Strength | Baseline
  Handgrip strength will be measured using a digital dynamometer to assess upper extremity muscle strength and overall muscular function.
Participant Satisfaction | Baseline
  Participant satisfaction with conventional and mixed reality-based assessments will be evaluated using a 10-point numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Zehra KORKUT, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Gülşah ÖZSOY, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Mehmet A GÜLER, PhD, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Yasemin GEDİKLİ ERTÜRK, MSc. in PT, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; İhsan KODAK, Assist. Prof. Dr., Study Chair — Kırşehir Ahi Evran University, School of Physical Therapy and Rehabilitation, Kırşehir, Türkiye; Haluk GÜMÜŞ, Prof. Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Süeda E YILMAZ, Dr., Study Chair — Rize State Hospital, Department of Neurology, Rize, Türkiye; Leyla ÖZTÜRK SÖNMEZ, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Tuğbanur BAYTOK, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye
Locations (1):
- Selcuk University Faculty of Medicine Hospital MS Life Center, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramari C, Hvid LG, David AC, Dalgas U. The importance of lower-extremity muscle strength for lower-limb functional capacity in multiple sclerosis: Systematic review. Ann Phys Rehabil Med. 2020 Mar;63(2):123-137. doi: 10.1016/j.rehab.2019.11.005. Epub 2019 Dec 6. PMID 31816449
- [Background] Casuso-Holgado MJ, Martin-Valero R, Carazo AF, Medrano-Sanchez EM, Cortes-Vega MD, Montero-Bancalero FJ. Effectiveness of virtual reality training for balance and gait rehabilitation in people with multiple sclerosis: a systematic review and meta-analysis. Clin Rehabil. 2018 Sep;32(9):1220-1234. doi: 10.1177/0269215518768084. Epub 2018 Apr 13. PMID 29651873
- [Background] Maggio MG, Russo M, Cuzzola MF, Destro M, La Rosa G, Molonia F, Bramanti P, Lombardo G, De Luca R, Calabro RS. Virtual reality in multiple sclerosis rehabilitation: A review on cognitive and motor outcomes. J Clin Neurosci. 2019 Jul;65:106-111. doi: 10.1016/j.jocn.2019.03.017. Epub 2019 Mar 18. PMID 30898488
- [Background] Massetti T, Trevizan IL, Arab C, Favero FM, Ribeiro-Papa DC, de Mello Monteiro CB. Virtual reality in multiple sclerosis - A systematic review. Mult Scler Relat Disord. 2016 Jul;8:107-12. doi: 10.1016/j.msard.2016.05.014. Epub 2016 May 21. PMID 27456884